CLINICAL TRIAL: NCT00367328
Title: To Determine The Efficacy Of A 1320nm Nd: YAG Nonablative Laser For Treatment of Hidradenitis Suppurativa
Brief Title: To Determine the Efficacy of a Laser Device for the Treatment of Hidradenitis Suppurativa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated: recruiting or enrolling participants has halted.
Sponsor: University of California, Davis (Other)
Collaborators: CoolTouch, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200513081-1
Record Dates: First submitted 2006-08-19; First posted 2006-08-22 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Supperativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): Oral Antibiotics in standard care vs. Laser treatment
  Interventions: Device: 1320nm Nd: YAG nonablative laser

INTERVENTIONS:
Device: 1320nm Nd: YAG nonablative laser — a 4 mm piece of skin tissue (about the size of a pencil-head eraser) from the affected area. This procedure is called a punch biopsy and will be done to confirm your diagnosis. A culture swab similar to a Q-Tip will be used to wipe the affected areas during the first visit to determine any bacteria that may be present. A survey with questions will be given at the first visit, again after 3 months and at the last visit to measure the success of the treatment. Photographs will be taken prior to each treatment and one month following your last treatment. A laser, which is a very powerful light, will be used to treat half of the skin that is affected by your condition.
  Other Names: laser treatment

SUMMARY:
A research study to determine the efficacy of a 1320 nm laser device for the treatment of hidradenitis suppurativa.

DETAILED DESCRIPTION:
Hidradenitis Suppurativa is a chronic, scarring disease. The treatments available for this condition are not very effective and work only for some patients.

Recently, a 1320nm laser device has been approved by the FDA for the treatment of acne and facial rejuvenation. Given the positive results seen with the use of this laser in the treatment of acne it is reasonable to hypothesize that a similar effect may be seen with the treatment of Hidradenitis suppurativa.

The specific aim of the study is to determine the efficacy of this device for the treatment of hidradenitis suppurativa as it relates to the patient's established treatment.

The investigators are trying to determine the efficacy of a laser for the treatment of hidradenitis suppurativa.

Patients will:

* be examined and interviewed
* have photographs taken of the treatment site
* have a 4mm punch biopsy performed
* have wound culture swabs performed

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* General good health and willingness to participate and ability to comply with the study protocol
* Biopsy proven hidradenitis suppurativa

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Hx of collagen vascular or photosensitive disorders
* Inability to follow-up with treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
A successful treatment is expected to improve the quality of life significantly by causing remission of disease. The data obtained from this study will also allow the development of laser-based treatment protocols for hidradenitis suppurativa. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical